CLINICAL TRIAL: NCT02180126
Title: Differing Levels of Positive Anti-Neutrophil Cytoplasm Antibody (ANCA) Test and Their Correlation With Vasculitis or Malignancy or Chronic Inflammation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC0041-14
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Positive ANCA: Patients with borderline positive ANCA results.
  Interventions: Other: Follow-up

INTERVENTIONS:
Other: Follow-up — Follow-up of of patients with borderline positive ANCA test results

SUMMARY:
A positive Anti-Neutrophil Cytoplasm Antibody (ANCA) test administered to patients with a high probability for vasculitis has high sensitivity and specificity for vasculitis. A positive ANCA test result in those patients who do not have a high probability for vasculitis requires extensive follow-up because those patients eventually present with malignancy or other inflammatory diseases. The investigators wish to investigate the correlation between the differing levels of positive ANCA tests and their relationship to vasculitis, malignancy and inflammatory diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with borderline positive ANCA test results

Exclusion Criteria:

* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with borderline positive ANCA test results who had been hospitalized at the Hillel Yaffe Medical Center.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Borderline Positive ANCA | Two weeks
  Borderline positive ANCA results of 12-19 U/ml is indication of possible malignancy or inflammatory diseases

CONTACTS AND LOCATIONS:
Overall Officials: Nina Avshovich, MD, Study Director — Hillel Yaffe Medical Center; Tatiana Sivan, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel